CLINICAL TRIAL: NCT06106802
Title: Lazertinib and Tepotinib for EGFR Mutant NSCLC in MET Overexpressed or Amplified Who Progressed After Lazertinib Treatment: A Phase II Multi-center Trial
Brief Title: Lazertinib & Tepotinib for EGFR Mutant NSCLC in MET Overexpressed or Amplified Who Progressed After Lazertinib Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, M.D. Professor, Division of hematology-oncology, Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-10-053
Record Dates: First submitted 2023-10-12; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — lazertinib; tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Patients will be treated with Lazertinib + tepotinib based on the MET FISH results.
  Lazertinib 240mg daily Tepotinib 500mg daily
  Interventions: Drug: Lazertinib; Drug: Tepotinib

INTERVENTIONS:
Drug: Lazertinib — Lazertinib 240mg/day
Drug: Tepotinib — Tepotinib 500mg/day

SUMMARY:
As the 3rd generation, EGFR TKI has become a standard treatment option for the 1st line therapy in EGFR mutated patients, the necessity for evaluating resistant mechanism to determine the matched subsequent therapeutic option has been highlighted. From the 1st line Osimertinib treatment, the heterogenous resistance mechanism has been observed showing most commonly by MET amplification (7-15%) followed by additional on-target EGFR mutation (6-10%), BRAF, PI3KCA, KRAS, HER2 mutation (13-14%) and still 40 to 50% remain unknown for the mechanism. (A. Leonetti et al.British Journal of Cancer(2019))

Based on the observation showing the MET amplification as the most common resistance mechanism to the 3rd generation EGFR TKI treatment, the "TATTON" study, a multi-arm, phase IB trial, demonstrated early clinical data of Osimertinib in combined with savolitinib. Among the patients, c-MET amplified patients who were previously treated with 3rd generation EGFR TKI, a combination of Osimertinib and savolitinib, showed an objective response rate of 33% and median PFS of 5.5 months. (G. Oxnard et al. Annals of Oncology(2020))

The clinical efficacy of Osimertinib with savolitinib in MET overexpressed or amplification patients are reported from the global phase II, "SAVANNAH" study. The preliminary results from the SAVANNAH trial showed that Osimertinib plus savolitinib demonstrated an objective response rate of 49% in patients with a high level of MET overexpression and/or amplification, defined as IHC90+ and/or FISH 10+, whose disease progressed on treatment with Osimertinib. The highest ORR was observed in patients with a high level of MET who were not treated with prior chemotherapy (52%). In patients whose tumors did not show a high level of MET, the ORR was 9% (MJ Ahn, WCLC, 2022). There are ongoing global Phase III SAFFRON study to validate the outcome from SAVANNAH study.

It has been reported that around 62% of tumor in Osimertinib progressed sample has MET overexpression and/or amplification, and more than one-third (34%) met the defined high MET level cut-off.

As Lazertinib is about to be approved as the treatment option for the treatment naïve EGFR mutated NSCLC, it is also becoming important to develop a further treatment plan based on the MET amplification status. In this study, the investigators designed a phase II study based on the MET amplification status to evaluate the clinical efficacy of Lazertinib + tepotinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed locally advanced or metastatic non-small cell lung cancer which is not amenable to treatment with a curative aim (e.g., surgery or radiation)
2. Confirmed EGFR mutations (exon 19 deletion, L858R) with acquired resistance after first-line lazertinib treatment (either partial response, complete response or stable disease last more than 6 months after initiation of Lazertinib) - patient can maintain the treatment with prior EGFR treatment as beyond progression until the patient start the treatment per this protocol
3. First-line cytotoxic chemotherapy received as palliative treatment is acceptable after the failure of Lazertinib (Patients with disease progression after adjuvant or neoadjuvant chemotherapy within 6 months are eligible to participate)
4. Patient with MET amplification FISH GCN ≥5 and/or MET/CEP7 ≥ 2 (If additional resistance mechanism to lazertinib, such as C797S, is observed with MET amplification, the recruitment needs to be discussed in advance with the principal investigator)
5. Available tissue for MET FISH
6. Age of 19 or more
7. Performance status of Eastern Cooperative Oncology Group 0 to 2
8. Expected minimum life expectancy of 12 weeks
9. Adequate organ function

   1. Absolute neutrophil count (ANC) ≥1500cells/mm3
   2. Platelet count ≥100,000cells/mm3
   3. Total bilirubin ≤1.5 x upper limit of normal(ULN)
   4. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN (or ≤5.0 x ULN, if liver metastasis is present)
   5. Creatinine level ≤1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 45mL/min (Calculated with Cockcroft- Gault equation)
10. Available to provide the adequate tissue and blood for the genomic tests

    - At least 20 unstained slide and 20 cc of blood at baseline and disease progression (If not, participant must be confirmed by the principal investigator
11. Agreed to perform re-biopsy at the timepoint of disease progression
12. Female subjects must either be of non-reproductive potential
13. Subject willing and able to comply with the protocol
14. Signed written informed consent

Exclusion Criteria:

1. Previously treatment with any kind of EGFR TKI other than lazertinib
2. All concurrent and/or other active malignant tumors requiring systemic therapy within 2 years prior to the initial administration of the investigational drug (However, the patient may participate if previous malignant tumor has been cured, and no further treatment is required)
3. Uncontrolled central nervous system metastases
4. Spinal cord compression, leptomeningeal carcinomatosis
5. Uncontrolled systemic illness, including uncontrolled hypertension, active bleeding, or active infection
6. Radiotherapy with a wide field of radiation within 2 weeks or radiotherapy with a limited field of radiation (localized radiotherapy or gamma knife surgery) for palliation within 1 week
7. Any unresolved toxicities from prior therapy, greater than CTCAE grade 1
8. Prior history of interstitial lung disease (ILD) or ILD like symptoms
9. Mean QT interval corrected for heart rate (QTc) ≥ 470 ms
10. No measurable lesion
11. Unable to swallow the product due to refractory nausea, vomiting or chronic gastrointestinal disease

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-02-02 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 9 months after completion of enrollment

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 60 months
Duration of Response (DoR) | up to 60 months
Disease control rate (DCR) | up to 60 months
Overall survival (OS) | up to 60 months

OTHER OUTCOMES:
Resistance mechanism analysis -tumor tissue | up to 60 months
  Using cf DNA acquired from baseline and at the time point of drug resistance, resistance mechanism will be evaluated. Using clinical outcome and confirmed mutation profile, resistance mechanism will be evaluated. Correlation between tissue and cfDNA based mutation profile will be analzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, Gangnam-gu, South Korea